CLINICAL TRIAL: NCT04484012
Title: A Phase 2 Study to Evaluate CD19-Specific Chimeric Antigen Receptor (CAR)-T Cells Combined With Acalabrutinib for Patients With Relapsed or Refractory Mantle Cell Lymphoma (MCL)
Brief Title: Modified Immune Cells (CD19 CAR T Cells) and Acalabrutinib for the Treatment of Relapsed or Refractory Mantle Cell Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19405; NCI-2020-04550 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 19405 (Other: City of Hope Comprehensive Cancer Center); P30CA033572 (NIH)
Record Dates: First submitted 2020-07-07; First posted 2020-07-23 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Recurrent Mantle Cell Lymphoma; Refractory Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — acalabrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (CD19 CAR T cells, acalabrutinib) (Experimental): Patients receive acalabrutinib PO BID on days -5 to 28 of cycle 1 and on days 1-28 of subsequent cycles. Patients also receive CD19 CAR T cells IV on day 0. Treatment with acalabrutinib repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients who have not attained CR after the first disease assessment and tolerated the initial CAR T cell infusion may receive a second CAR T cell infusion in cycle 2.
  Interventions: Drug: Acalabrutinib; Biological: CD19CAR-CD28-CD3zeta-EGFRt-expressing Tn/mem-enriched T-lymphocytes

INTERVENTIONS:
Drug: Acalabrutinib — Given PO
  Other Names: ACP-196; Bruton Tyrosine Kinase Inhibitor ACP-196; Calquence
Biological: CD19CAR-CD28-CD3zeta-EGFRt-expressing Tn/mem-enriched T-lymphocytes — Given IV
  Other Names: CD19CAR-CD28-CD3zeta-EGFRt-expressing Tn/mem-enriched T Cells; CD19R(EQ)28zeta/EGFRt+ Naive and Memory T Cells; CD19R(EQ)28zetaEGFRt+ Tn/mem Cells

SUMMARY:
This phase II trial investigates the side effects of CD19 chimeric antigen receptor (CAR) T cells and acalabrutinib, and to see how well they work in treating patients with mantle cell lymphoma that has come back (relapsed) or does not respond to treatment (refractory). T cells are infection fighting blood cells that can kill cancer cells. The T cells given in this study will come from the patient and will have a new gene put in them that makes them able to recognize CD19, a protein on the surface of the cancer cells. These CD19-specific T cells may help the body's immune system identify and kill CD19 positive cancer cells. Acalabrutinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving CD19 CAR T cells together with acalabrutinib may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the safety of adding CD19CAR-CD28-CD3zeta-EGFRt-expressing Tn/mem-enriched T-lymphocytes (CD19 CAR T cells) to acalabrutinib treatment. (Safety Lead-in) II. Estimate the complete response (CR) rate within 6 months after adding CD19 CAR T cells to acalabrutinib treatment. (Phase 2)

SECONDARY OBJECTIVES:

I. Assess best response, time to and duration of CR. II. Estimate the 1-year progression free survival (PFS) rate and overall survival (OS).

III. Describe the full toxicity profile.

EXPLORATORY OBJECTIVES:

I. Assess CD19-CAR T cell persistence. II. Assess CD19-CAR T cell activity as measured by CD19 B cell aplasia. III. Describe the duration of CR from completion of acalabrutinib. IV. Describe immunogenicity of CD19-CAR T cells in the presence of the BTK inhibitor.

V. Characterize CD19 expression on tumor cells. VI. Describe cytokine profile after CD19-CAR T cell infusion. VII. Determine BTK and PLCG2 mutational status prior to treatment.

OUTLINE:

Patients receive acalabrutinib orally (PO) twice daily (BID) on days -5 to 28 of cycle 1 and on days 1-28 of subsequent cycles. Patients also receive CD19 CAR T cells intravenously (IV) on day 0. Treatment with acalabrutinib repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients who have not attained CR after the first disease assessment and tolerated the initial CAR T cell infusion may receive a second CAR T cell infusion in cycle 2.

After completion of study treatment, patients are followed up at 3, 6 and 12 months, then yearly for up to 15 years post CAR T cells infusion.

ELIGIBILITY:
Inclusion Criteria Informed Consent and Willingness to Participate

1. All participants must have the ability to understand and the willingness to sign a written informed consent.
2. Participants must agree to allow the use of archival tissue from diagnostic tumor biopsies.

   * If unavailable, exceptions may be granted with Study PI approval. Note: For research participants who do not speak English, a short form consent may be used with a COH certified interpreter/translator to proceed with screening and leukapheresis, while the request for a translated full consent is processed.

   Age Criteria
3. Age 18 years and older. Performance Status
4. ECOG Performance status ≤ 2 or KPS ≥ 70% (Appendix A) Nature of Illness and Treatment-Related Criteria
5. Documented CD19+ MCL by flow cytometry or IHC (from biopsy) if prior CD19 directed therapy was previously used

   a. BM is optional at enrollment IF patient already has biopsy proven disease.
6. Participants must be currently receiving acalabrutinib and have been taking acalabrutinib for between 3 and 7 months prior to initiating screening procedures on the study and:

   1. must have at least 1 prior regimen (not including single-agent corticosteroids)
   2. best response to acalabrutinib therapy is MRD+ CR, PR or SD at the time of screening b (1) must have measurable disease by CT scan (≥ 1.5 cm) or evidence of blood, spleen, skin, gastrointestinal (GI) or bone marrow involvement Note: Participants who are on other BTK inhibitors, but will thereafter be switched to acalabrutinib prior to lymphodepletion, may be eligible provided that the duration of all BTK inhibitor therapy was ≤ 3-7 months
7. No contraindications to leukapheresis, steroids or tocilizumab Clinical Laboratory Criteria (To be performed within 28 days prior to enrollment)
8. Total serum bilirubin ≤ 2.0 mg/dL Participants with Gilbert syndrome may be included if their total bilirubin is ≥ 3.0 x ULN and direct bilirubin ≤ 1.5 x ULN.
9. Blood counts:

   * Absolute Neutrophil count (ANC ≥1000 cells/ul)*

     * Growth factor use within 7 days prior screening is not allowed
   * Platelet count ≥75,000/ul. Transfusion with 7 days prior to screening is not allowed* *Exception: participants with bone marrow involvement do not need to meet this criteria
10. AST < 3 x ULN
11. ALT < 3 x ULN
12. Creatinine clearance of ≥ 50 mL/min per the Cockcroft-Gault formula
13. International Normalized Ratio (INR) OR Prothrombin (PT) ≤ 1.5 x ULN
14. Activated Partial Thromboplastin Time (aPTT) ≤ 1.5 x ULN
15. Female of childbearing potential: negative urine or serum pregnancy test. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
16. Cardiac function (12 lead-ECG): QTc must be ≤ 480 msec
17. Left ventricular ejection fraction >40%
18. Oxygen saturation 92% or above at room air or DLCO of 40% of best predicted Contraception
19. Participants of reproductive potential must agree to use highly effective birth control methods throughout therapy and for 2 months after final CAR T cell infusion and/or 2 days after final acalabrutinib dose, whichever is later (See Section 5.12 and Appendix B).

Exclusion Criteria Previous therapies

1. Allogeneic hematopoietic cell transplantation (HCT) within the last 6 months.
2. Autologous HCT within the last 3 months.
3. Prior failure of any BTK inhibitor therapy. (Participant WILL be allowed if, after administration of other BTK inhibitors they have switched to acalabrutinib prior to lymphodepletion, and if the duration of all BTK inhibitor therapy was ≤ 3-7 months).
4. Participants known to have mutations associated with resistance to BTK inhibitors from prior studies.

   Concomitant therapies
5. Concurrent use of systemic steroids or chronic use of immunosuppressant medications. Recent or current use of inhaled steroids is not exclusionary. Physiologic replacement of steroids (i.e., prednisone ≤ 7.5 mg /day, or hydrocortisone ≤ 20 mg /day) is allowed. During study participation, participants may receive systemic corticosteroids as needed for treatment-emergent comorbid conditions.
6. Approved anti-cancer therapies other than acalabrutinib are not allowed after enrollment, with the exception of steroids or involved field radiation to control progressive disease during cell manufacturing, prior to lymphodepletion/start of protocol therapy.
7. Requires treatment with a strong cytochrome P450 3A4 (CYP3A4) inhibitor/inducer.
8. Unable to discontinue anticoagulation with warfarin or equivalent vitamin K antagonists (e.g., phenprocoumon) within 7 days of leukapheresis and remain off through end of study treatment.

   Other illnesses or conditions
9. Class III/IV cardiovascular disability according to the New York Heart Association Classification. Subjects with controlled, asymptomatic atrial fibrillation can enroll.
10. Participants with clinically significant arrhythmia or arrhythmias not stable on medical management.
11. Active auto-immune disease requiring systemic immunosuppressive therapy, including uncontrolled autoimmune hemolytic anemia (AIHA) or idiopathic thrombocytopenic purpura (ITP).
12. Suspected or confirmed progressive multifocal leukoencephalopathy (PML).
13. Requires major surgical procedure within 28 days prior to first dose of study drug. If a subject has major surgery, they must have recovered adequately from any toxicity and/or complications from the intervention before the first dose of study drug.
14. Participants with a known history or prior diagnosis of optic neuritis or other immunologic or inflammatory disease affecting the central nervous system.
15. Known history of drug-specific hypersensitivity or anaphylaxis to either study agent.
16. Malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel that is likely to affect absorption, symptomatic inflammatory bowel disease, partial or complete bowel obstruction, or gastric restrictions and bariatric surgery, such as gastric bypass.
17. Known bleeding disorders (e.g., von Willebrand's disease or hemophilia)
18. History of stroke or intracranial hemorrhage within 6 months prior to enrollment.
19. History of other malignancies, except for the following: malignancy surgically resected (or treated with other modalities) with curative intent, adequately treated in situ carcinoma of the breast or cervix uteri, basal cell carcinoma of the skin or localized squamous cell carcinoma of the skin; early stage prostate cancer on expectant management; malignancy treated with curative intent with no known active disease present for ≥ 3 years.
20. Lactating women.
21. Active chronic graft-versus-host disease (GVHD) post-allogeneic HCT.
22. Uncontrolled active infection:

    * HIV positive or have active hepatitis B or C infection based on testing performed within 4 weeks of enrollment.
    * Hepatitis B or C serologic status: subjects who are hepatitis B core antibody (anti-HBc) positive and who are surface antigen negative will need to have a negative polymerase chain reaction (PCR) result. Those who are hepatitis B surface antigen (HbsAg) positive or hepatitis B PCR positive will be excluded.
    * Subjects who are hepatitis B core antibody positive (or have a known history of HBV infection) should be monitored quarterly with a quantitative PCR test for HBV DNA. HBV monitoring should last until 12 months after last dose of study drug. Any subject with a rising viral load (above lower limit of detection) should discontinue study drug and have antiviral therapy instituted and a consultation with a physician with expertise in managing hepatitis B. Subjects who are core Ab positive at study enrollment are strongly recommended to start Entecavir before start and until completion of study treatment.
    * Subjects who are hepatitis C antibody positive will need to have a negative PCR result. Those who are hepatitis C PCR positive will be excluded.
    * Subjects who are positive cytomegalovirus [CMV] DNA polymerase chain reaction [PCR]).
    * Subject with any active significant bacterial, fungal or viral (other than those listed) infections.
23. Any other condition that would, in the Investigator's judgment, contraindicate the subject's participation in the clinical study due to safety concerns with clinical study procedures.

    Noncompliance
24. Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics).

    * Eligibility should be confirmed per institutional policies.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2020-12-31 (Actual); Primary Completion 2026-09-02 (Estimated); Study Completion 2026-09-02 (Estimated)

PRIMARY OUTCOMES:
Occurrence of dose-limiting toxicities (DLTs) (Safety Lead-in) | Day 0 up to 28 days after the first chimeric antigen receptor (CAR) T cell infusion
  Rates and associated 95% Clopper and Pearson exact confidence interval (CI) will be estimated for DLTs at the safe dose.
Complete response (CR) (Phase II) | Within 6 months of CAR T-cell infusion and concurrent acalabrutinib therapy
  Response will be assessed based on Lugano classification. CR rate is defined as the proportion of response-evaluable participants who achieve a best response of CR within 6 months of CAR T-cell infusion and concurrent acalabrutinib therapy. Rates and associated 95% Clopper and Pearson exact CI will be estimated for CR within 6 months.

SECONDARY OUTCOMES:
Time to CR | From the first achievement of CR after CAR T cell infusion through disease relapse or progression or death, assessed up to 15 years
  Descriptive statistics will be used to summarize the time to CR among those who achieve CR.
Duration of CR | From the first achievement of CR after CAR T cell infusion through disease relapse or progression or death, assessed up to 15 years
  Duration of CR will be assessed using Kaplan Meier methods.
Best response | Up to 1 year post CAR T cell infusion
  Defined as the best response documented at any time after CAR T cell infusion through 1 year after CAR T cell infusion or the start of any non-protocol anti-lymphoma therapy, whichever occurs first. Best response will be presented in tabular format including counts and percentages.
Progression-free survival (PFS) | From start of protocol treatment (start of lymphodepletion) to the first observation of disease relapse/progression or death due to any cause, whichever occurs first, assessed at 1 year
  Progression-free survival will be assessed using Kaplan Meier methods.
Overall survival (OS) | From start of protocol treatment (start of lymphodepletion) to death due to any cause, assessed at 1 year
  OS will be assessed using Kaplan Meier methods.
Incidence of adverse events | Up to 15 year post CAR T cell infusion
  Toxicities will be recorded using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5. Observed toxicities will be summarized by type, severity, date of onset (per each treatment cycle or follow-up period), and attribution.

OTHER OUTCOMES:
CD19 CAR T cell persistence | At 28 days
  Rates and associated 95% Clopper and Pearson exact CI will be estimated for CD19 CAR T cell persistence at 28 days.
Presence of CD19CAR immunogenicity | Up to 1 year post CAR T cell infusion
  Rates and associated 95% Clopper and Pearson exact CI will be estimated for presence of CD19CAR immunogenicity.
Duration of CR from completion of acalabrutinib | Up to 15 years post CAR T cell infusion
  This analysis will include only participants who have achieved CR and completed 6 cycles of acalabrutinib, and it will be defined as the time from last dose of acalabrutinib through disease relapse, progression or death, whichever is earlier. Will be assessed using Kaplan Meier methods.

CONTACTS AND LOCATIONS:
Overall Officials: Lihua E Budde, Principal Investigator — City of Hope Comprehensive Cancer Center
Locations (1):
- City of Hope Comprehensive Cancer Center, Duarte, California, United States